CLINICAL TRIAL: NCT02085928
Title: Clinical and Ultrasonographic Results of Intratissue Percutaneous Electrolysis (EPI Technique) in Chronic Lateral Epicondylitis: a Case Series With Prospective 12 Months Follow up
Brief Title: Clinical and Ultrasonographic Results of Intratissue Percutaneous Electrolysis in Lateral Epicondylitis
Status: Completed | Type: Observational
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Other Study IDs: CEU-005
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Lateral Epicondylitis
Keywords: Tennis elbow; Lateral epicondylitis; Intratissue percutaneous electrolysis; Eccentric exercise; Ultrasonography
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lateral epicondylitis: Patients with lateral epicondylitis with persistent pain for at least 3 months
  Interventions: Other: Intratissue percutaneous electrolysis, associated with eccentric exercise and stretching

INTERVENTIONS:
Other: Intratissue percutaneous electrolysis, associated with eccentric exercise and stretching — * The EPI technique was performed under ultrasound-guidance on the clinically relevant area (or areas of maximum tenderness to palpation and with ultrasonographic degenerative tendon changes) using an intensity of 4-6 mA during 3 seconds, approximately 3 times. We used the EPI machine (Cesmar Electromedicina S.L., Barcelona, Spain) and a GE Logiq E Portable Ultrasound Machine with GE Linear probe 12L-RS (5-13 mhz) (GE Healthcare, Wisconsin, EEUU).
  * The eccentric exercise program consisted of three series of up to 10 repetitions of eccentric work, repeated twice daily (morning and afternoon), under maximum load (initially with one kilogram) in an optimal and functional pain-free range.
  * The stretching program consisted of a stretching exercise for the epicondylar muscles consisting in three series of 7 repetitions twice a day (morning and afternoon.

SUMMARY:
Lateral epicondylitis (LE) is the most common cause of lateral elbow pain. Intratissue percutaneous electrolysis (EPI technique) is a novel minimally invasive approach which consists in the application of a galvanic current through a puncture needle which produces a local inflammatory process in the soft tissue and the reparation of the affected tissue.

The purpose of this study is to evaluate the clinical and ultrasonographic effectiveness of a multimodal program using the intratissue percutaneous electrolysis technique and exercises in the short term for patients with chronic lateral epicondylitis, and to determine whether the clinical outcomes achieved decline over time.

This study is an observational one-way repeated measures design. 36 patients in a clinical setting presenting with lateral epicondylitis (mean age = 38, mean time since injury = 12.6 months) received one session of EPI per week over 4-6 weeks, associated with a home program of eccentric exercise and stretching. The main outcome measures were severity of pain (VAS, digital algometer, Cozen and Thompson tests), disability (DASH questionnaire), structural tendon changes (ultrasound), hypervascularity (power doppler) and patient's perceptions of overall outcome (4-point scale). Measurements at 6, 26 and 52 weeks follow-up included recurrence rates (increase of severity of pain or disability compared to discharge), the perception of overall outcome and success rates. Paired Student t-tests and Chi squared tests were applied to data. Enrollment into this study ended in September 2012.

All outcome measures registered significant improvements between pre-intervention and discharge. Most patients (30, i.e. 83.3%) rated overall outcome as 'successful' at 6 weeks. The ultrasonographic finding revealed that the hypoechoic regions and hypervascularity of the extensor carpi radialis brevis change significantly. At 26 and 52 weeks, all participants (32) perceived a 'successful' outcome. Recurrence rates were null after discharge, and at the 6, 26 and 52 week follow-ups.

DETAILED DESCRIPTION:
Patients received one session of EPI technique per week over 4 weeks (or over 6 weeks when pain persisted) associated with a home program consisting of eccentric exercise (EccEx) and stretching, initiated 24 hours after each session. The EccEx and stretching program was taught by a physiotherapist in the first session and monitored in subsequent sessions. At discharge, patients were instructed to perform only EccEx once daily for the first 6 weeks of the follow-up period.

The EPI technique was performed under ultrasound-guidance on the clinically relevant area (or areas of maximum tenderness to palpation and with ultrasonographic degenerative tendon changes) using an intensity of 4-6 milliampere (mA) during 3 seconds, approximately 3 times. The investigators used the EPI machine (Cesmar Electromedicina S.L., Barcelona, Spain) and a GE Logiq E Portable Ultrasound Machine with GE Linear probe 12L-RS (5-13 mhz) (GE Healthcare, Wisconsin, EEUU). During the EPI technique, the patient was placed in a supine position, with the affected elbow placed in a position of 90° flexion and maximum pronation. The elbow was sterilized and the sonographic transducer, enclosed in a sterile cover over sterile applied gel, was placed at the lateral epicondyle (first approach) and over the humeroradial joint between the head of the radius and the capitulum of the humerus (second approach), where it remained throughout the procedure. A common target area was the deep surface of the common extensor tendon (origin of the ECRB [extensor carpi radialis brevis] and the EDC [extensor digitorum communis]) (first approach) and the deep surface of the ECRB, over the capsule and the lateral ulnar collateral ligament (second approach). A 0.3 x 25mm. (1 inch) needle was inserted at a 30° to 45° angle to the skin in the direction of the lateral epicondyle (first approach) and at a 80° angle to the skin, with the needle tip directed towards the humeroradial joint (second approach). In the first approach the needle was advanced parallel to the longitudinal plane of the tendon (in-plane approach); whereas in the second approach the needle was advanced along the short plane of the humeroradial joint (out-of-plane approach). Real-time ultrasonographic imaging provided guidance for both procedures. Once the needle reached the target tissue, readjustments of the needle position were made in order to ensure a correct stimulation. The generation of the galvanic current creates a white image (hyperechoic) as a result of the liberation of hydrogen gas due to the electrolysis. Oral paracetamol was used when necessary for the purpose of pain relief only.

The eccentric exercise program consisted of three series of up to 10 repetitions of eccentric work, repeated twice daily (morning and afternoon), under maximum load (initially with one kilogram) in an optimal and functional pain-free range. From maximum wrist extension and radial deviation, rapid wrist flexion movement were performed, followed by a 2-second hold of the final position. In between series patients were given a rest period of 2-3 minutes. This formula was used for the duration of the physiotherapy program. The concentric contraction phase for returning to the starting position was nullified with the help of the other hand.

The stretching program consisted of a stretching exercise for the epicondylar muscles consisting in three series of 7 repetitions twice a day (morning and afternoon), performed in a sitting position with a flexed wrist and fingers, ulnar deviation and elbow extension reaching the stretch limit without bounces, and held for 45 seconds, with a 30-second rest between repetitions.

ELIGIBILITY:
Individuals who meet all of the following criteria are eligible for enrollment into the study:

Inclusion Criteria:

* Adult between 18-45 years of age
* Pain over the lateral humeral epicondyle provoked by at least two of the following: gripping, palpation, stretching of forearm extensor muscles and resisted wrist or middle finger extension
* Persistent pain for at least 3 months despite conservative treatments including medication (oral nonsteroidal antiinflammatory drugs (NSAIDs) and analgesics), brace application, or physiotherapy
* Patients with structural tendon changes at the origin of the extensors, demonstrated during musculoskeletal ultrasound

Individuals who meet any of the following criteria are disqualified from enrollment of the study:

Exclusion Criteria:

* Patients with a history of advanced cervical arthrosis in the C4-C6 segments.
* Bilateral LE with central sensitization
* Symptoms compatible with posterior interosseous nerve entrapment.
* Previous surgery, fractures, trauma or previous history of rheumatic disorders in the area of the lateral epicondyle
* History of corticosteroid injection at the lateral epicondyle within the last 3 months

Two experienced professionals performed recruitment and examination of subjects in order to assess for eligibility criteria. All eligible patients provided written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 36 participants with lateral epicondylitis
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain at treatment discharge and at 6 weeks. | Baseline, at treatment discharge and at 6 weeks.
  * Intensity of elbow pain during activity was recorded using a visual analogue scale (VAS) score (0=no pain; 100=maximum intensity).
  * Pain-free pressure was measured with a digital algometer (Wenzhou Sundoo Instruments Co., Ltd, China).
  * Cozen and Thompson tests were performed in order to provoke localized pain over the lateral epicondyle.

SECONDARY OUTCOMES:
Change from baseline in disability at treatment discharge and at 6 weeks. | Baseline, at treatment discharge and at 6 weeks.
  - Disability was measured with the DASH questionnaire (0-100, being 100 the higher disability).
Change from baseline in ultrasound imaging at treatment discharge and at 6 weeks. | Baseline, at treatment discharge and at 6 weeks.
  - Structural tendon changes were examined in the lateral epicondylar area, including the origin of the extensor tendon, ECRB, and the adjacent soft tissues with a GE Logiq E Portable Ultrasound Machine (GE Healthcare, Wisconsin, EEUU) under the guidelines defined by the European Society of Musculoskeletal Radiology. Structural tendon changes (tendon thickening, hypoechogenicity and intrasubstance tears) were demonstrated by the grey-scale US, and hypervascularity (not present or several areas) by Power Doppler (PD) examination. The same experienced professional performed all US and PD examinations and was blinded as to the phase of treatment.
Change from at treatment discharge in recurrence at 6 weeks. | At treatment discharge, 6 weeks.
  - Success rates were then calculated based on perception of overall outcome; we considered excellent or good to be 'successful' and fair or poor to 'unsuccessful'
Change from 6 weeks in recurrence at 26 and 52 weeks. | 6 weeks, 26 weeks and 52 weeks.
  - Success rates were then calculated based on perception of overall outcome; we considered excellent or good to be 'successful' and fair or poor to 'unsuccessful'
Change from at treatment discharge in patient's perceptions of overall outcome, at 6 weeks. | At treatment discharge, 6 weeks.
  - We also measured patient's perceptions of overall outcome using a 4-point scale: 'excellent' in the case of full return to all activity with no pain, 'good' if full return to all activity occurred with occasional mild pain, 'fair' if no pain was present with normal activities but significant pain occurred with heavy activities; and 'poor' in the case of little or no relief of pre-operative symptoms)
Change from 6 weeks in patient's perceptions of overall outcome, at 26 and 52 weeks. | 6 weeks, 26 weeks, and 52 weeks.
  - We also measured patient's perceptions of overall outcome using a 4-point scale: 'excellent' in the case of full return to all activity with no pain, 'good' if full return to all activity occurred with occasional mild pain, 'fair' if no pain was present with normal activities but significant pain occurred with heavy activities; and 'poor' in the case of little or no relief of pre-operative symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Fermin Valera-Garrido, PT, PhD, Principal Investigator — CEU San Pablo University; MVClinic
Locations (1):
- CEU San Pablo University, Boadilla del Monte, Madrid, Spain

REFERENCES:
- [Derived] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629